CLINICAL TRIAL: NCT01420250
Title: Phase I Trial of Weekly Cabazitaxel With Concurrent Intensity Modulated Radiation Therapy and Androgen Deprivation Therapy for the Treatment of Locally Advanced High Risk Adenocarcinoma of the Prostate
Brief Title: Cabazitaxel With Radiation and Hormone Therapy for Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11D.243; 2011-32 (Other: CCRRC); JT 1820 (Other: JeffTrial Number)
Record Dates: First submitted 2011-08-17; First posted 2011-08-19 (Estimated); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Adenocarcinoma of the prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — cabazitaxel; XRP6258; Radiotherapy, Intensity-Modulated; Radiotherapy; bicalutamide; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Cabazitaxel with Intensity Modulated Radiation Therapy (IMRT) (Experimental): Weekly Cabazitaxel with concurrent IMRT
  Interventions: Drug: Cabazitaxel; Radiation: Intensity Modulated Radiation Therapy (IMRT); Drug: Anti-Androgen Therapy: Bicalutamide; Genetic: Luteinizing Hormone-Releasing Hormone (LHRH) Agonist

INTERVENTIONS:
Drug: Cabazitaxel — Administered weekly on the same day of radiation according to the following infusion levels:
  Level 1 (Initial): 4 mg/m2; Level -1: 2 mg/m2; Level 2: 6 mg/m2; Level 3: 8 mg/m2; Level 4: 10 mg/2;
  Other Names: Jevtana; XRP-6258
Radiation: Intensity Modulated Radiation Therapy (IMRT) — Starts 8 weeks after initiation of androgen deprivation therapy, given daily at 1.8 Gy for a total of 75.6 Gy
  Other Names: Intensity Modulated Radiation Therapy; IMRT; Radiation therapy
Drug: Anti-Androgen Therapy: Bicalutamide — * Taken once daily by mouth starting between 2 weeks and 1 day before the first administration of Luteinizing Hormone-Releasing Hormone (LHRH)
  * Will continue once daily until the final day of IMRT
  Other Names: Casodex; Cosudex; Calutide; Kalumid
Genetic: Luteinizing Hormone-Releasing Hormone (LHRH) Agonist — * First administration will occur 1 day to 2 weeks after the start of Bicalutamide and 8 weeks prior to the start of IMRT (+/- 4 weeks)
  * Will continue for 24 months after IMRT
  * Total administered duration and agent used must be documented on the case report form
  Other Names: Gonadotropin-releasing hormone; GnRH; LHRH; Luliberin

SUMMARY:
This is a single-center, open-label, non-randomized Phase I study of weekly Cabazitaxel with concurrent intensity modulated radiation therapy (IMRT) (A type of 3-dimensional radiation therapy that uses computer-generated images to show the size and shape of the tumor. Thin beams of radiation of different intensities are aimed at the tumor from many angles.) and androgen deprivation therapy (Treatment to suppress or block the production or action of male hormones) in patients with locally advanced prostate cancer.

It is hoped that by adding Cabazitaxel to the standard IMRT, greater local disease control can be achieved and eventually the cure rate can be increased. After this study, the maximally tolerated dose of Cabazitaxel that could be used in combination with radiation can be found.

Men with locally advanced high risk prostate cancer represent a group of patients for whom cure is potentially achievable utilizing a multimodality approach. More aggressive treatment upfront with chemotherapy and ADT may improve the long term disease control. We hypothesize that Cabazitaxel may be added to radiation therapy safely, and we anticipate that this novel approach will improve disease control and eventually improve survival for locally advanced prostate cancer patients.

DETAILED DESCRIPTION:
Patients with locally advanced high Gleason grade prostate cancer often have local and metastatic disease progression. To improve on these outcomes, therapy needs to be directed at controlling the androgen sensitive and insensitive prostate cancer cells in the primary and metastatic sites. This therapeutic challenge has further prompted the use of combined modality approaches incorporating chemotherapy and hormonal therapy with radiation aimed at the intrinsically resistant cells and the micrometastatic disease that are both androgen sensitive and resistant. High likelihood of occult metastatic disease and existence of intrinsically castration resistant cells are the main rationales for early institution of androgen deprivation therapy (ADT) and chemotherapy in prostate cancer.

The rationale for combining chemotherapeutic agents with ADT and radiotherapy in high risk prostate cancer patients is based on that chemotherapy can enhance radiotherapy and is also an effective therapy for metastatic castrate resistant disease. Prior studies with weekly docetaxel with ADT and intensity modulated radiation therapy (IMRT) were safe and feasible however cabazitaxel is more potent mitotic inhibitor which may further enhance the outcomes of patients with locally advanced prostate cancer.

Men with locally advanced high risk prostate cancer represent a group of patients for whom cure is potentially achievable utilizing a multimodality approach. More aggressive treatment upfront with chemotherapy and ADT would improve the long term disease control. We hypothesize that Cabazitaxel may be added to radiation therapy safely, and we anticipate that this novel approach will improve disease control and eventually improve survival for locally advanced prostate cancer patients.

The safety of the combination of Cabazitaxel with radiation will be established after this study. Potential efficacy will be determined in the future phase II/III trials. Hypofraction radiation treatment with shorter duration maybe possible if combined with chemotherapy modality.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of the prostate with locally advanced prostate cancer without distant metastatic with unfavorable risk features that are defined below:
* Gleason score ≥8
* Gleason score 7 and T3/T4 disease
* Gleason score 7 but PSA ≥20
* Karnofsky Performance Status >70,
* Age > 18
* Performance Status: ECOG ≤2
* Peripheral neuropathy: must be < grade 1
* Hematologic (minimal values):
* Absolute neutrophil count > 1,500/mm3
* Hemoglobin > 8.0 g/dl
* Platelet count > 100,000/mm3
* Hepatic function
* Total bilirubin < Upper limit of normal (ULN)(except for Gilbert's disease)
* AST (SGOT) < 1.5 x ULN
* ALT (SGPT) < 1.5 x ULN
* Creatinine < 1.5 x ULN
* Men of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter.
* No history of previous chemotherapy or pelvic irradiation

Exclusion Criteria:

* Patients with a history of severe hypersensitivity reaction to Cabazitaxel or other drugs formulated with polysorbate 80.
* History of urological surgery or procedures predisposing to GU complications after radiation (will be determined by radiation oncologist)
* History of diverticulitis, rectal bleeding or other lower GI diseases predisposing to GI complications after radiation (will be determined by radiation oncologist)
* History of prior chemotherapy or pelvic irradiation,
* History of prior invasive malignant cancer(s) within the last 5 years except adequately treated or controlled basal cell or squamous cell carcinoma of the skin
* Documented distant metastatic disease.
* Prior radical prostatectomy or cryosurgery for prostate cancer or bilateral orchiectomy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-09-22 (Actual); Primary Completion 2015-07-21 (Actual); Study Completion 2020-07-21 (Actual)

PRIMARY OUTCOMES:
Maximally Tolerated Dose (MTD) of Cabazitaxel and Intensity Modulated Radiation Therapy (IMRT) | Weekly during treatment then every 3 months until 2 years after completion of IMRT
  To determine the maximally tolerated dose, or the safety and feasibility, of the concurrent weekly Cabazitaxel and IMRT with androgen deprivation therapy

SECONDARY OUTCOMES:
Acute and Late Non-Hematologic and Hematologic Toxicity Profile of Cabazitaxel and Intensity Modulated Radiation Therapy (IMRT) Combination | Weekly during IMRT, then at 2 weeks and 3 months after IMRT, and then every 3 months until 2 years after IMRT
  The toxicity profile will be recorded according to the NCI CTCAE v4.0 criteria. Toxicity assessment will be performed weekly during IMRT, then at 2 weeks and 3 months after IMRT, and then every 3 months until 2 years after IMRT.
5-Year Biochemical Relapse Free Survival | Within 5 years after completion of IMRT
  A PSA rise by 2 ng/mL or more above the nadir PSA is considered as biochemical relapse after external beam IMRT (ASTRO 2005 Phoenix criteria).

CONTACTS AND LOCATIONS:
Overall Officials: Robert Den, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Thomas Jefferson University Hospitals — http://www.JeffersonHospital.org/